CLINICAL TRIAL: NCT04351984
Title: Transcatheter Mitral Valvuloplasty for Severe Mitral Regurgitation Pilot Study
Brief Title: Transcatheter Mitral Valvuloplasty Pilot Study
Acronym: MitraClip
Status: Completed | Type: Observational
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Associate Professor, Division of Cardiology, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2020-04
Record Dates: First submitted 2020-04-16; First posted 2020-04-17 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Mitral Valve Insufficiency; Mitral Regurgitation; Mitral Valve Regurgitation
Keywords: MitraClip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Mitral Regurgitation
  Interventions: Device: MitraClip

INTERVENTIONS:
Device: MitraClip — Transcatheter Mitral Valvuloplasty with MitraClip
  Other Names: Transcatheter Mitral Valvuloplasty

SUMMARY:
This study is to evaluate the efficacy and safety of Transcatheter Mitral Valvuloplasty for Severe Mitral Regurgitation

ELIGIBILITY:
Inclusion Criteria:

* Significant symptomatic mitral regurgitation (MR ≥ 3+) due to primary abnormality of the mitral apparatus [degenerative MR] in patients who have been determined to be at prohibitive risk for mitral valve surgery by a heart team, which includes a cardiac surgeon experienced in mitral valve surgery and a cardiologist experienced in mitral valve disease, and in whom existing comorbidities would not preclude the expected benefit from reduction of the mitral regurgitation.
* Age 19 and more
* Written informed consent

Exclusion Criteria:

* Patients who cannot tolerate procedural anticoagulation or post-procedural antiplatelet regimen
* Active endocarditis of the mitral valve
* Rheumatic mitral valve disease
* Evidence of intracardiac, inferior vena cava (IVC) or femoral venous thrombus

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe mitral regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mitral regurgitation | 1 month

SECONDARY OUTCOMES:
All cause death | 1 year
Stroke | 1 year
Myocardial infarction | 1 year
Re-hospitalization | 1 year
Acute kidney dysfunction | 5 days
Vascular complication | 5 days
Bleeding | 5 days
Successful valvuloplasty | 5 days
  No significant complication

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided